CLINICAL TRIAL: NCT06214195
Title: Clinical Study on the Use of Shengmai San to Prevent Anthracycline Sequential Trastuzumab Therapy Related Cardiac Toxicity
Brief Title: The Use of Shengmai San to Prevent Anthracycline Sequential Trastuzumab Therapy Related Cardiac Toxicity
Acronym: START
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Huang Ping, Associate chief physician, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZCHBC025
Record Dates: First submitted 2023-11-25; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Cardiotoxicity Induced by Drug Therapy for Breast Cancer
Keywords: prevent; cardiotoxicity; trastuzumab; chemotherapy; anthracycline
MeSH Terms: conditions — Cardiotoxicity | interventions — fructus schizandrae, radix ginseng, radix ophiopogonis drug combination; schizandrin

STUDY DESIGN:
Intervention Model Description: The risk exposure factors for the experimental group and the control group are the same
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): Provide preventive treatment with Shengmai San
  Interventions: Drug: Shengmai San (ingredients include ginseng, Ophiopogon japonicus, and Schisandra chinensis)
- control group (No Intervention): No preventive intervention

INTERVENTIONS:
Drug: Shengmai San (ingredients include ginseng, Ophiopogon japonicus, and Schisandra chinensis) — Ginseng 6g , Ophiopogon japonicus 12g ,Schisandra chinensis 5g , other secondary Chinese medicines can be added according to the doctor's judgment and the patient's condition，decoction in water, one dose and two decoctions, taken twice a day, continuously for 7 days from the start of each chemotherapy cycle (± 3 days), including anthracyclines and taxanes (the frequency and dosage of medication can be adjusted according to adverse reactions in the later stage); The total duration of medication interventionis 7 days per cycle, with a total of 8 cycles. If the chemotherapy is less than 8 cycles, continue taking for 7 consecutive days from the start of each subsequent trastuzumab cycle (the frequency and dosage can be adjusted based on adverse reactions) until a total of 8 cycles are reached.
  Arms: treatment group

SUMMARY:
To evaluate the effectiveness and safety of Shengmai San in preventing anthracycline sequential trastuzumab therapy related cardiac toxicity through a prospective randomized controlled study.

DETAILED DESCRIPTION:
This study is a randomized, controlled, open-label prospective clinical study. This study adopts an optimal design, with the main evaluation indicator being the incidence of cardiac toxicity. Patients who passed the inclusion and exclusion criteria through clinical research were randomly assigned to the experimental group and control group. Experimental(treatment)group: received preventive treatment with Shengmai Powder，and may also receive additional Chinese medicines based on the doctor's judgment and the patient's condition.Control group: during chemotherapy and trastuzumab administration, no Chinese medicine with ginseng, ophiopogon japonicus and schisandra chinensis as ingredients or western medicine with heart strengthening or heart protection function were used. During the treatment process, cardiac function related indicators such as symptomatic congestive heart failure or asymptomatic but decreased left ventricular ejection fraction (LVEF) are evaluated to determine the occurrence of cardiac toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Non metastatic primary invasive HER2 positive breast cancer stage I-III invasive HER2 positive breast cancer is defined as the tumor invasive component HER2 immunohistochemical IHC+++or IHC++confirmed to be HER2 positive by fluorescence in situ hybridization
2. Plan to use AC sequential TH (P) adjuvant or neoadjuvant chemotherapy with anthracycline containing chemotherapy regimens (A is doxorubicin or epirubicin, C is cyclophosphamide, T is paclitaxel, liposome paclitaxel, albumin bound paclitaxel or docetaxel, H is trastuzumab, which can be combined with pertuzumab (P))，and before using anthracycline drugs, the left ventricular ejection fraction (LVEF) should be ≥ 50%
3. Plan to use trastuzumab or trastuzumab combined with pertuzumab for one year of treatment；
4. ECOG PS: 0-1 points；
5. The patient has good compliance with the planned treatment and follow-up, can understand the research process of this study, and sign a written informed consent form.

Exclusion Criteria:

1. The New York Heart Association (NYHA) classifies patients with heart disease at or above Level II (including Level II)
2. Severe heart disease or discomfort, including high-risk uncontrolled arrhythmia, etc
3. There are contraindications or intolerance to treatment with trastuzumab, including allergies to trastuzumab, and the presence of underlying heart diseases that cannot be treated with trastuzumab as determined by a specialist
4. Previously allergic to ginseng, Ophiopogon japonicus, and Schisandra chinensis
5. Unable to cooperate with treatment and follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2024-01-20 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of cardiotoxicity in the treatment group and control group | From 1 week before enrollment to 1.5 years after the start of trastuzumab treatment.
  Calculate the incidence of cardiotoxicity associated with anthracycline sequential trastuzumab treatment of two groups.Cardiotoxicity is defined as the occurrence of symptomatic congestive heart failure, or a decrease in left ventricular ejection fraction (LVEF) without clinical symptoms that meets one of the following conditions: ① a decrease of ≥ 15% in LVEF from baseline after anti-cancer treatment; ② After anti-cancer treatment, LVEF decreased by ≥ 10% from baseline and the monitoring value was<50%; ③ LVEF monitoring value after anti-cancer treatment is less than 45%. The definition of symptomatic congestive heart failure includes but is not limited to any one or more of the following: moist rales in the lungs, anterior tibial edema in both lower limbs, and cyanosis of the lips.

SECONDARY OUTCOMES:
The incidence of adverse events in the treatment group and control group, except for cardiotoxicity | From the use of anthracycline drugs or Shengmai San to 1.5 years after the start of trastuzumab treatment.
  Using the Common Terminology Criteria for Adverse Events (CTC AE) version 5.0, evaluate the adverse events and toxic reactions of the two groups, except for cardiotoxicity, to determine the incidence rate.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Huang, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Can apply to researchers

REFERENCES:
- [Background] Eiermann W; International Herceptin Study Group. Trastuzumab combined with chemotherapy for the treatment of HER2-positive metastatic breast cancer: pivotal trial data. Ann Oncol. 2001;12 Suppl 1:S57-62. PMID 11521723
- [Background] Seidman A, Hudis C, Pierri MK, Shak S, Paton V, Ashby M, Murphy M, Stewart SJ, Keefe D. Cardiac dysfunction in the trastuzumab clinical trials experience. J Clin Oncol. 2002 Mar 1;20(5):1215-21. doi: 10.1200/JCO.2002.20.5.1215. PMID 11870163
- [Background] Farolfi A, Melegari E, Aquilina M, Scarpi E, Ibrahim T, Maltoni R, Sarti S, Cecconetto L, Pietri E, Ferrario C, Fedeli A, Faedi M, Nanni O, Frassineti GL, Amadori D, Rocca A. Trastuzumab-induced cardiotoxicity in early breast cancer patients: a retrospective study of possible risk and protective factors. Heart. 2013 May;99(9):634-9. doi: 10.1136/heartjnl-2012-303151. Epub 2013 Jan 24. PMID 23349345